CLINICAL TRIAL: NCT02032966
Title: Outcomes Following Surgical Versus Nonsurgical Treatment of Fibular Fractures Following Operative Fixation of Unstable Medial Malleolus Fractures: A Prospective Randomized Study
Brief Title: Surgical Versus Nonsurgical Treatment of Fibular Fractures: A Prospective Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Collaborators: Southeastern Fracture Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-010
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Ankle Fracture; Malleolus Fracture; Medial Malleolus Fracture; Bimalleolar Fracture; Trimalleolar Fracture
Keywords: outcomes; surgical; non-surgical; ankle; malleolus; fracture; tibia; fibula; bimalleolar; trimalleolar
MeSH Terms: conditions — Ankle Fractures; Fractures, Bone | interventions — Periodontal Debridement; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nonsurgical (Experimental): Randomized to "nonsurgical": patient will receive surgical treatment of the inside portion (medial malleolus) of the tibia fracture only; the fibula fracture (and posterior malleolus fracture, if present) will be closed reduced (not repaired surgically).
  Interventions: Procedure: Nonsurgical
- Surgical (Active Comparator): Randomized to "surgical": patient will receive surgical treatment of both the inside portion (medial malleolus) of the tibia fracture, as well as the fibula fracture (lateral malleolus). Fixation of the posterior side of the tibia (posterior malleolus) may or may not be performed based upon intraoperative x-rays.
  Interventions: Procedure: Surgical
- syndesmotic injury (Other): Non-randomized / "syndesmotic injury": patients who have a positive ligament stress test (signifying a syndesmotic injury) during surgery will require surgical treatment of both the tibia and the fibula and cannot be randomized to either arm ("nonsurgical" versus "surgical"). Patients in this arm will still be included in the study for the collection of clinical and functional outcomes.
  Interventions: Procedure: Surgical

INTERVENTIONS:
Procedure: Nonsurgical — Randomized to "nonsurgical": patient will receive surgical treatment of the inside portion (medial malleolus) of the tibia fracture only; the fibula fracture (and posterior malleolus fracture, if present) will be closed reduced (not repaired surgically).
  Arms: Nonsurgical
Procedure: Surgical — Randomized to "surgical": patient will receive surgical treatment of both the inside portion (medial malleolus) of the tibia fracture, as well as the fibula fracture (lateral malleolus). Fixation of the posterior side of the tibia (posterior malleolus) may or may not be performed based upon intraoperative x-rays.
  Arms: Surgical; syndesmotic injury

SUMMARY:
Isolated surgical repair of the inside portion of the tibia may be enough to stabilize an ankle fracture in which both the tibia and the fibula are broken. This would alleviate the need for another incision, plate, and screws to repair the fibula. The purpose of this study is to help determine if surgically repairing only the tibia fracture will lead to equivalent clinical outcomes when compared with surgical repair of both bones.

The hypothesis of this study is that operative stabilization of the medial malleolus fracture only, in otherwise ligamentously stable bimalleolar and/or trimalleolar fractures of the ankle, will lead to equivalent clinical outcomes and functional scores as those treated with operative stabilization of both malleoli and/or all malleoli.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients ≥ 18 years of age with acute, closed bimalleolar and/or trimalleolar ankle fractures
* Operative fixation of the ankle fracture is within 3 weeks from date of injury
* Bimalleolar and/or trimalleolar ankle fractures in which the medial malleolus fragment is greater than 1.7cm wide on lateral x-ray imaging
* Bimalleolar and/or trimalleolar ankle fractures in which the posterior malleolus fragment is less than 20% of the depth of the tibial articular surface

Exclusion Criteria:

* Skeletally immature patients < 18 years of age
* Single malleolar ankle fractures
* Open fractures
* Operative fixation of the ankle fracture is more than 3 weeks from date of injury
* Bimalleolar and/or trimalleolar fractures in which the medial malleolar fragment is less than or equal to 1.7cm wide on lateral x-ray imaging
* Bimalleolar and/or trimalleolar ankle fractures in which the posterior malleolus fragment is greater than or equal to 20% of the depth of the tibial articular surface
* Ankles with previous fractures of the medial and/or lateral malleolus requiring operative intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
clinical outcomes | one year
  Time to union (radiographic healing of the fracture), Time to weight-bearing, Complications

SECONDARY OUTCOMES:
functional outcomes | one year
  Measured by the SF-36 Health Survey and the Foot Function Index

CONTACTS AND LOCATIONS:
Overall Officials: Dirk W Kiner, M.D., Principal Investigator — UTCOM Chattanooga/Erlanger Health System
Locations (1):
- Erlanger Health System, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No